CLINICAL TRIAL: NCT05017766
Title: NCCR AntiResist: Mono-center Study to Identify New Approaches to Combat Antibiotic-resistant Bacteria.
Brief Title: NCCR AntiResist:: New Approaches to Combat Antibiotic-resistant Bacteria
Acronym: AntiResist
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02588; pe20Khanna
Record Dates: First submitted 2021-07-26; First posted 2021-08-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Antimicrobial Resistance (AMR)
Keywords: National Center of Competence in Research (NCCR); Urinary tract infection (UTI); Pneumonia; Deep-seated infections; E. coli; Klebsiella species; S. aureus; P. aeruginosa; bacterial properties; Community-acquired pneumonia (CAP); Hospital-acquired pneumonia (HAP); Ventilator-associated pneumonia (VAP); cystic fibrosis (CF)
MeSH Terms: conditions — Urinary Tract Infections; Pneumonia; Escherichia coli Infections; Klebsiella Infections; Staphylococcal Infections; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual samples from routinely collected material (urine, tracheal secretion in intubated patients, sputum in cystic fibrosis patients, bronchoalveolar lavage fluid, blood, deep-seated infectious material that is surgically removed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- A) Urinary tract infection: Processing of residual urine for proteomic, metabolomic and transcriptomic analysis, immunocytochemical or fluorescence in-situ hybridisation (FISH) analysis, flow cytometry analysis (FACS), immunophenotyping. If positive for target bacteria: sample stored at biobank. If previous antibiotic treatment: plasma sample storage. Exploration of bacterial properties (Highly sensitive mass spectrometry, whole genome sequencing), expression of virulence factors, genomic alterations of bacterial species, metabolism, surface molecule expression, gene expression levels, cytokine levels, immune cell biology, antibiotic concentration (chromatography/mass spectrometry). Demographical, clinical, microbiological, laboratory, epidemiological and hospital-associated data will be analysed. 500 samples per target bacteria (S. aureus, P. aeruginosa, E. coli, Klebsiella species) included. First, a pilot study from randomly selected patients within each bacterial species group (n=50, each) is done.
  Interventions: Other: analysis of antimicrobial resistance
- B) Pneumonia: Processing of residual samples (tracheal secretion, bronchioalveolar lavage (BAL)) for proteomic, metabolomic, transcriptomic and cytological analysis. If positive for target bacteria: sample stored at biobank. If previous antibiotic treatment: plasma sample storage. Exploration of bacterial properties. Demographical, clinical, microbiological, laboratory, epidemiological and hospital-associated data will be analysed. 500 samples per target bacteria (S. aureus, P. aeruginosa, E. coli, Klebsiella species) included.
  Interventions: Other: analysis of antimicrobial resistance
- C) Deep-seated infections: Processing of intraoperative material residual samples for proteomic, metabolomic, transcriptomic and cytological analysis. If positive for target bacteria: sample stored at biobank. Exploration of bacterial properties. Demographical, clinical, microbiological, laboratory, epidemiological and hospital-associated data will be analysed. 500 samples per target bacteria (S. aureus, P. aeruginosa, E. coli, Klebsiella species) included.
  Interventions: Other: analysis of antimicrobial resistance
- D) Controls for A), B) and C): Control samples result from patients with a suspected infection (infection sites A), B) or C), in which no microbiological confirmed infection has been diagnosed. Storage at biobank
  Interventions: Other: analysis of antimicrobial resistance
- E) Clinical controls for A), B) and C) without obtained samples: For clinical controls, clinical characteristics of patients with detection of target pathogens in their routine samples (but which could not be included for sample analysis in this study) will be assessed.
  Interventions: Other: analysis of antimicrobial resistance
- F) Cohort with analysis whether the application of Article (Art) 34 HFV can avoid a bias: Since part of the data and samples in this study are collected with the representative consent of the ethics committees, it is investigated whether the application of Art. 34 HFV prevents selection bias with respect to the study population. For this purpose, differences between the actual study population using Art. 34 HFV and the study population with provided research consent will be descriptively investigated in terms of the prevalence of multi-resistant germs and other available population characteristics.
  Interventions: Other: analysis of antimicrobial resistance

INTERVENTIONS:
Other: analysis of antimicrobial resistance — In samples from patients infected with one of the focus pathogens (E. coli, Klebsiella species, S. aureus, P. aeruginosa) will be:
  (i) isolated and pathogenic bacteria characterized; (ii) pathogen in-situ properties at single-cell and bulk average determined; (iii) human metabolites, proteins and cells determined (iv) antibiotic concentration determined (v) bacterial growth monitored
  Deducted from the data will be:
  1. relevant human components and pathogen properties that are common to most patients with similar indication
  2. underlying regulatory networks and triggers in pathogen cells and human tissues.
  Clinical outcomes (survival/mortality) and treatment response (response or failure) will be correlated to the in vitro retrieved host and bacterial data.

SUMMARY:
This is an explorative, mono-center study including prospectively collected patient samples from the University Hospital of Basel. It is to investigate antimicrobial resistance (AMR) including three clinical manifestations of infectious diseases: urinary tract infection, pneumonia and deep-seated infections. The focus is on four bacteria (E. coli, Klebsiella species, S. aureus, P. aeruginosa) that are part of the high priority list of World Health Organization (WHO). Residual patient samples are analysed for proteomic, metabolomic and transcriptomic analysis, immunocytochemical or fluorescence in-situ hybridisation (FISH) analysis, flow cytometry analysis (FACS) and immunophenotyping and exploration of bacterial properties.

DETAILED DESCRIPTION:
The National Center of Competence in Research (NCCR) AntiResist aims at utilizing patient samples in order to investigate the physiology of bacterial pathogens in human patients and establishing a unique multidisciplinary network of clinicians, biologists, engineers, chemists, computational scientists and drug developers.

The goal of this project is to elucidate the physiological properties of bacterial pathogens in infected human patients in order to provide new ways of combatting superbugs. These clinical data will be used to guide and benchmark development of patient-mimicking and in-vitro models, accelerate the search for novel bacterial targets, antibacterial compounds and non-conventional strategies.

In detail, the focus will be on three clinical manifestations of infectious diseases caused by four critical bacterial pathogens belonging to WHO "priority pathogens" list: E. coli, Klebsiella species, S. aureus and P. aeruginosa :

A) Urinary tract infection B) Pneumonia C) Deep-seated infections D) Controls for A), B) and C) E) Clinical controls for A), B) and C) without obtained samples F) Analysis whether the application of Art. 34 HFV (Weiterverwendung biologischen Materials und/oder gesundheitsbezogener Personendaten für die Forschung bei fehlender Einwilligung und Information) can avoid a bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed (i) urinary tract infection, (ii) pneumonia (including patients after lung transplantation, cystic fibrosis) or (iii) deep-seated infection with focus pathogen:

  * E. coli
  * Klebsiella species
  * S. aureus
  * P. aeruginosa
* Controls: no detectable bacteria in routine microbiology lab and no other infection site at inclusion of the sample and follow up for 10 days, signed general consent
* Clinical controls without obtained samples, but with confirmed (i) urinary tract infection, (ii) pneumonia (including patients after lung transplantation, cystic fibrosis) or (iii) deep-seated infection with focus pathogen:

  * E. coli
  * Klebsiella species
  * S. aureus
  * P. aeruginosa

Exclusion Criteria:

* Patients who have refused research and reuse of their data/samples (e.g. general consent) or any other decline (e.g. Patientenverfügung).
* other than one of the focus bacteria in routine microbiology lab
* Age: <18 years
* Controls without signed general consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient samples during routine collection at the University Hospital of Basel from November 2020 to approximately December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome: survival rate | one time assessment at baseline
  Survival rate (correlated to the in vitro retrieved host and bacterial data. In vitro retrieved host and bacterial data include: Proteomics, Metabolomics, FISH, Histology, PCR/Microbial genome sequencing, Microbial transcriptome, Antibiotic concentration, Timelapse studies, phenotypic characterisations, molecular typing, innate immune response characterization, Antibiotic tolerance testing, Microfluidic systems, 3-D models, Transcriptomics, Flow cytometry (FACS))
Clinical outcome: mortality rate | one time assessment at baseline
  Mortality rate (correlated to the in vitro retrieved host and bacterial data. In vitro retrieved host and bacterial data include: Proteomics, Metabolomics, FISH, Histology, PCR/Microbial genome sequencing, Microbial transcriptome, Antibiotic concentration, Timelapse studies, phenotypic characterisations, molecular typing, innate immune response characterization, Antibiotic tolerance testing, Microfluidic systems, 3-D models, Transcriptomics, Flow cytometry (FACS))
Treatment response (binary: yes/ no) | one time assessment at baseline
  Treatment response (correlated to the in vitro retrieved host and bacterial data. In vitro retrieved host and bacterial data include: Proteomics, Metabolomics, FISH, Histology, PCR/Microbial genome sequencing, Microbial transcriptome, Antibiotic concentration, Timelapse studies, phenotypic characterisations, molecular typing, innate immune response characterization, Antibiotic tolerance testing, Microfluidic systems, 3-D models, Transcriptomics, Flow cytometry (FACS))

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Prof., Principal Investigator — University Hospital Basel, Division of Infectiology
Locations (1):
- University Hospital Basel, Basel, Switzerland